CLINICAL TRIAL: NCT03979157
Title: Non-invasive Molecular Imaging to Determine Hemoglobin and Collagen Levels in Muscles Before and After Exercise, and Over Time
Brief Title: Non-invasive Molecular Imaging of Muscle Structure (MSOT_muscles)
Acronym: MSOT_muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 169_19B
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Muscular Diseases
Keywords: Muscular Diseases; Duchenne muscular disease; MSOT
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Multispectral Optoacoustic Tomography (MSOT) of proximal and distal leg muscles (total of 12 sites: left and right, 3 measurement points of Musculus quadriceps, and 3 measurement points of Musculus triceps surae) before and after the 6-Minute-Walk-Test by to independent investigators. Repetition of the same protocol after 14 days.
  Interventions: Device: Multispectral Optoacoustic Tomography

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography — Non-invasive transcutaneous imaging of subcellular muscle components

SUMMARY:
This study aims to determine hemoglobin and collagen levels in muscles before and after exercise, and over time, using Multispectral Optoacoustic Tomography (MSOT). During MSOT, a transducer is placed on the skin similar to a conventional sonography and instead of sound, energy is supplied to the tissue by means of light flashes. This leads to a constant change of minimal expansions and contractions (thermoelastic expansion) of individual tissue constituents or molecules. The resulting sound waves can then be detected by the same examination unit.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is one of the most common progressive childhood muscle diseases with an incidence of 1 in 3500 male newborns and is associated primarily with decreased life expectancy. Pathogenetically, there is a deficiency of dystrophin, a structural protein of the sarcolemma, which is caused by mutations (usually deletions) of the dystrophin gene (Xp21.3-p21.2). The result of dystrophin deficiency is a necrosis of muscle cells that are replaced by connective tissue and adipose tissue. Clinical scores (6-minute walk test, 6MWT) and MRI studies to characterize the degenerative changes of skeletal muscle in the early stages are available for the quantitative assessment of the disease progression as well as therapy effects, the significance of which is controversially discussed. However, the highly sensitive assessment of gene therapy effects will become increasingly important in the future. Sensitive, non-invasive methods for the detection of early muscle degeneration and muscle function in the course are of great clinical and scientific importance.

MSOT has already been demonstrated to be a potential monitoring tool in different diseases. However, it has not yet been investigated to what extent 1) previous physical activity 2) different measuring ranges at the muscle, 3) longitudinal measurements and 4) intra- and interoperative variability influences the measured results. In particular, molecular changes immediately after the 6-MWT are relevant for studies in patients with DMD.

In this first pilot study, the investigators want to investigate in healthy adults, whether increased exercise changes the hemoglobin values, whether the collagen content remains constant and whether repeated measurements at different muscle positions by different investigators provide consistent results over time. This information is indispensable for future studies of children with muscular diseases in order to be able to make statements about disease progression or even therapy response.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age

Exclusion Criteria:

* any reference to a myopathy
* pregnancy
* tattoo in the scanning region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Muscular collagen content | one time point ( 2 measurements on day 1)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers compared before and after 6-MWT.
Muscular myo-/hemoglobin content | one time point ( 2 measurements on day 1)
  Quantitative myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers compared before and after 6-MWT.

SECONDARY OUTCOMES:
Muscular oxygenated and deoxygenated myo-/hemoglobin content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative oxygenated and deoxygenated myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers compared before and after 6-MWT and after 14 days.
Intraindividual collagen content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) compared between three different points in one muscle of one healthy volunteer
Intraindividual myo-/hemoglobin content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) compared between three different points in one muscle of one healthy volunteer
Intraindividual oxygenated and deoxygenated myo-/hemoglobin content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative oxygenated and deoxygenated myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) compared between three different points in one muscle of one healthy volunteer
Muscular collagen content in men and women | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative collagen signal of muscles derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in healthy men compared to healthy women.
Muscular myo-/hemoglobin content in men and women | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative myo-/hemoglobin signal of muscles derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in healthy men compared to healthy women.
Muscular oxygenated and deoxygenated myo-/hemoglobin content in men and women | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative oxygenated and deoxygenated myo-/hemoglobin signal of muscles derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in healthy men compared to healthy women.
Correlation of collagen signal with the 6-MWT | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in Healthy volunteers before and after exercise correlated with the 6-MWT
Correlation of myo-/hemoglobin signal with the 6-MWT | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in Healthy volunteers before and after exercise correlated with the 6-MWT
Correlation of oxygenated and deoxygenated myo-/hemoglobin signal with the 6-MWT | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative oxygenated and deoxygenated myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in Healthy volunteers before and after exercise correlated with the 6-MWT
Interrater reliability of collagen content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers before and after 6-MWT and after 14 days compared between to investigators
Interrater reliability of myo-/hemoglobin content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers before and after 6-MWT and after 14 days compared between to investigators
Interrater reliability of oxygenated and deoxygenated myo-/hemoglobin content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative oxygenated and deoxygenated myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers before and after 6-MWT and after 14 days compared between to investigators
Interreader reliability of collagen content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers before and after 6-MWT and after 14 days compared between to readers
Interreader reliability of myo-/hemoglobin content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers before and after 6-MWT and after 14 days compared between to readers
Interreader reliability of oxygenated and deoxygenated myo-/hemoglobin content | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative oxygenated and deoxygenated myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers before and after 6-MWT and after 14 days compared between to readers
Muscular collagen content over time period | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers compared between day 1 and after 14 days.
Muscular myo-/hemoglobin content over time period | multiple time points ( 2 measurements on day 1 and 2 measurements on day 15)
  Quantitative myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in muscles of healthy volunteers compared between day 1 and after 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Regensburger, Dr., Principal Investigator — Department of Pediatrics and Adolescent Medicine, University of Erlangen; Ferdinand Knieling, Dr., Principal Investigator — Department of Pediatrics and Adolescent Medicine, University of Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request as follows:
  * Individual participant data will not be available
  * Study Protocol and Statistical Analysis Plan will be available
  * The data will be available beginning 9 months and ending 36 months following article publication.
  * The data will be available to researchers who provide a methodologically sound proposal.
  * The data will be available for individual participant data for meta-analysis, only.
  * Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at https://www.uk-erlangen.de.
  Restrictions may apply due to patient privacy and the General Data Protection Regulation.
Supporting Information: Study Protocol, SAP
Time Frame: 36 months after publication
Access Criteria: Resonable request

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03979157/SAP_000.pdf
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03979157/Prot_001.pdf